CLINICAL TRIAL: NCT00237250
Title: Efficacy and Safety of Vildagliptin in Subjects With Impaired Glucose Tolerance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2357
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Prediabetic State
Keywords: Pre-diabetes; vildagliptin; IGT
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to placebo in lowering post-meal blood glucose levels in people with pre-diabetes who have high blood sugar levels after meals.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* Body mass index (BMI) in the range 23-45

Exclusion Criteria:

* Diagnosis of diabetes
* Serious cardiovascular events within the past 6 months
* Use of insulin or any oral antidiabetic agent
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change in area under the 0-2 hour prandial glucose curve at 12 weeks

SECONDARY OUTCOMES:
Adverse event profile after 12 weeks of treatment
Change in ratio for postprandial insulin AUC and postprandial glucose AUC (0-2 hours) after 12 weeks of treatment
Change in HOMA B at 12 weeks
Change in fasting insulin at 12 weeks
Change in fasting proinsulin/insulin ratio at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Rosenstock J, Foley JE, Rendell M, Landin-Olsson M, Holst JJ, Deacon CF, Rochotte E, Baron MA. Effects of the dipeptidyl peptidase-IV inhibitor vildagliptin on incretin hormones, islet function, and postprandial glycemia in subjects with impaired glucose tolerance. Diabetes Care. 2008 Jan;31(1):30-5. doi: 10.2337/dc07-1616. Epub 2007 Oct 18. PMID 17947341